CLINICAL TRIAL: NCT01072422
Title: Smoking Cessation in Primary Health Care Patients With Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Lena Lundh, RN MScN, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPN 2008/1929-31/5; HSN 0803-0374 (Other Grant/Funding Number: Stockholm County Council)
Record Dates: First submitted 2010-02-19; First posted 2010-02-22 (Estimated); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Smoking; Pulmonary Disease, Chronic Obstructive
Keywords: Smoking; Pulmonary Disease, Chronic Obstructive; Questionnaires; Nurses; Primary Health Care
MeSH Terms: conditions — Smoking; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- counseling based on answers in TTQ (Experimental): 40 participating primary health care nurses will be randomly assigned to this arm. Each nurse will identify 5 consecutive patients with COPD who smoke (n = 200 total patients). The nurses will ask the patients to fill in the assessment protocol, TTQ. The nurses will then provide an intervention to each patient in the form of individual treatment on the basis of that patient's answers to the TTQ.
  Interventions: Behavioral: smoking cessation

INTERVENTIONS:
Behavioral: smoking cessation — Use of trying to quit smoking instrument and quit smoking advice

SUMMARY:
The purpose of this study is to determine if an assessment protocol that measures the need for support with smoking cessation and that will be administered by primary health care nurses helps patients with obstructive pulmonary disease (COPD) quit smoking.

DETAILED DESCRIPTION:
Some patients with COPD continue to smoke despite the importance of quitting. A specially developed assessment protocol for such patients may support nurses in their discussions with the patients about smoking cessation. In a previous qualitative study involving in-depth interviews with patients with COPD, the assessment protocol "Trying to quit smoking" (TTQ) was developed. The protocol consists of approximately 21 statements that the patient responds to on a scale ranging from 1 (agree entirely) to 4 (disagree). The purpose of the protocol is to identify areas in which the patient may need extra support in order to quit smoking.

The aim of this study is to validate the TTQ by testing it in a clinical setting. The study will be conducted at approximately 40 primary health care centers in Stockholm County. The nurses will identify 5 consecutive patients who have COPD and smoke. All nurses will complete a questionnaire for each patient at baseline (after visit 1) and after 3 months describing treatment provided. The nurses will ask each patient to fill in the TTQ and will provide individual counseling on the basis of the answers. After 3 months, the nurses will ask all patients if they still smoke and to fill in the TTQ again. Appropriate statistical methods will be used to analyze the questionnaire data.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of COPD
* Current smoker
* Speak Swedish well enough to answer the TTQ assessment protocol

Exclusion Criteria:

* Cognitive difficulties that, in the judgment of the participating nurses, would make it difficult for the patient to answer the TTQ assessment protocol or benefit from counseling

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2010-03; Primary Completion 2013-04 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Smoking cessation | 3 months after patients' first visit to primary health care center

SECONDARY OUTCOMES:
Validity of protocol | Immediately after patients fill in protocol (baseline and 3 months after first visit to primary health care center)

CONTACTS AND LOCATIONS:
Overall Officials: Lena Lundh, MSc nursing, Principal Investigator — Karolinska Institutet
Locations (1):
- 200 primary health care centers across Stockholm County, Stockholm, Sweden